CLINICAL TRIAL: NCT00503854
Title: Fatigue and Symptom Burden in Febrile Neutropenia
Brief Title: Fatigue and Symptom Burden in Low-Risk Cancer Patients Undergoing Treatment for Febrile Neutropenia
Status: Completed | Type: Observational
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: 2005-0936; NCI-2018-02184 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2005-0936 (Other: M D Anderson Cancer Center); P30CA016672 (NIH)
Record Dates: First submitted 2007-07-17; First posted 2007-07-19 (Estimated); Last update posted 2018-10-22 (Actual); Status verified 2018-10

CONDITIONS: Fatigue; Febrile Neutropenia; Solid Neoplasm
MeSH Terms: conditions — Fatigue; Febrile Neutropenia | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Observational (questionnaire): Patients complete a questionnaire on days 1, 2, and 6 regarding fatigue, sleep disturbance, depression, and other symptoms.
  Interventions: Behavioral: Questionnaire

INTERVENTIONS:
Behavioral: Questionnaire — Ancillary studies
  Other Names: Questionnaires

SUMMARY:
This trial studies how fatigue and symptom burden in low-risk cancer patients undergoing treatment for febrile neutropenia. Cancer and numerous cancer treatments are associated with various symptoms including anemia, fever, and neutropenia, which may also be associated with fatigue. Treating low-risk cancer patients for febrile neutropenia may reduce levels of fatigue.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES I. To determine whether fatigue improves as patients are treated for febrile neutropenia (Day #1, Day #2 and Day #6).

SECONDARY OBJECTIVES I. To identify clinical factors associated in cancer patients with low risk for outpatient treatment of febrile neutropenia on either outpatient febrile neutropenia treatment pathway presenting with moderate to severe fatigue.

II. To describe demographic information in cancer patients with low risk for outpatient treatment of febrile neutropenia and fatigue while enrolled in either of two outpatient febrile neutropenia treatment pathways.

OUTLINE:

Patients complete a questionnaire on days 1, 2, and 6 regarding fatigue, sleep disturbance, depression, and other symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Cancer patients with solid tumors at low risk for outpatient treatment of febrile neutropenia evaluated in the EC and enrolled in outpatient febrile neutropenia pathways (pathway 1 or 2). Low risk is defined as hemodynamically stable solid tumor patients that do not have pneumonia or are on steroids. Febrile neutropenia is marked by a temperature greater than or equal to 38.3 degrees Celsius and an absolute neutrophil count (ANC) less than or equal to 1000 within 24 hours.
* Patients must be able to speak, read and write in English.
* Patients must be able to complete the required survey tools independently.
* Patients must report a moderate to severe fatigue level to question # 3 of the Brief Fatigue Inventory (BFI) (4 or greater on a 0-10 scale) on EC admission day.
* Pregnant women if they meet eligibility criteria of the febrile neutropenia (NF) pathway and are able to take the oral/intravenous (IV) antibiotic prescribed by the pathway.

Exclusion Criteria:

* Patients will be excluded from the study if they are not on the neutropenic pathway at the time of study entry.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Outpatient seen at MD Anderson Cancer Center
Sampling Method: Non-Probability Sample
Enrollment: 70 (Actual)
Dates: Start 2007-05-31 (Actual); Primary Completion 2018-04-05 (Actual); Study Completion 2018-04-05 (Actual)

PRIMARY OUTCOMES:
Mean fatigue level evaluated by Brief Fatigue Inventory (BFI) | Up to day 6
  Improvement in mean fatigue level will be assessed. Summary statistics, such as mean, standard deviation, median and range will be provided at the Emergency Center (EC) admission and along the treatment period at days 1, 2, and 6. Exploratory plots such as scatter plots and box plots will also be prepared. For those patients requiring longer time of treatment (greater than 7 days) and remaining on the febrile neutropenia (NF) pathway, the fatigue levels at the time of pathway discharge will also be summarized. The change in fatigue levels between day 1 and day 6 will be calculated for each item in the BFI. Wilcoxon signed rank test will be used to assess the significance of change. The change in fatigue score for question # 3 between EC admission and day 6 of the study will also be calculated and assessed using Wilcoxon signed rank test.

SECONDARY OUTCOMES:
Clinical factors associated with cancer patients with low risk for outpatient treatment of febrile neutropenia | Up to day 6
  Will be explored using descriptive statistics, bivariate correlation and scatter plots. The association between each clinical factor and fatigue improvement (yes or no) will be assessed using Wilcoxon's rank-sum test (for continuous clinical factors) or Pearson's chi^2 test (for categorical clinical factors). Univariate and multivariable logistic regression models will be fit using fatigue severity as a dependent variable and baseline demographic information, clinical factors and laboratory values as potential predictors. Anemia, using granulocyte-colony stimulating factor (G-CSF) before enrollment will be controlled for as confounding variables in the model. The goodness-of-fit of the model will be evaluated using partial residual plots. Furthermore, a multivariable linear mixed model will be fit for the repeating measurements of fatigue scores, which takes into account the correlation among the scores obtained within the same subject over time.
Demographic information in cancer patients with low risk for outpatient treatment of febrile neutropenia and fatigue | Up to day 6
  Will be explored using descriptive statistics, bivariate correlation and scatter plots. Univariate and multivariable logistic regression models will be fit using fatigue severity as a dependent variable and baseline demographic information, clinical factors and laboratory values as potential predictors. Furthermore, a multivariable linear mixed model will be fit for the repeating measurements of fatigue scores, which takes into account the correlation among the scores obtained within the same subject over time. The mixed model will include a random patient effect and baseline demographic information, clinical factors and laboratory values will be fit as fixed effects.

CONTACTS AND LOCATIONS:
Overall Officials: Carmen Escalante, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center Website — http://www.mdanderson.org